CLINICAL TRIAL: NCT04408313
Title: A Comparative Effectiveness Trial of Extended Release Naltrexone Versus Extended Release Buprenorphine With Individuals Leaving Jail
Brief Title: Extended Release Naltrexone Versus Extended Release Buprenorphine With Individuals Leaving Jail
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1UG1DA050077 (NIH)
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-02

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XR-B (Experimental): Extended-release buprenorphine
  Interventions: Drug: XR-B
- XR-NTX (Active Comparator): Extended-release naltrexone
  Interventions: Drug: XR-NTX

INTERVENTIONS:
Drug: XR-B — Individuals will receive extended-release buprenorphine, administered as a subcutaneous injection, is available in seven different dosage strengths for weekly (8, 16, 24, and 32 mg) and monthly (64, 96, and 128 mg) administration by a health care professional.
  Other Names: extended-release buprenorphine
  Arms: XR-B
Drug: XR-NTX — Injectable naltrexone will be used, at a dose of 4cc (380mg of naltrexone), administered by intramuscular injection to the buttocks (alternating sides monthly). Individuals will receive monthly injections.
  Other Names: extended-release naltrexone
  Arms: XR-NTX

SUMMARY:
The proposed study is a Type 1 hybrid effectiveness-implementation trial. Individuals with opioid use disorder in county jails throughout the state of Maryland will be randomly assigned within gender within jail to one of two groups: Arm 1. XR-B (n=120). XR-B in jail followed by 6 monthly injections post-release at a community treatment program. Arm 2. XR-NTX (n=120). One injection of XR-NTX in jail, followed by 6 monthly injections post-release at a community treatment program.

DETAILED DESCRIPTION:
This study is a Type 1 hybrid effectiveness-implementation trial. County jails willing to provide extended-release naltrexone (XR-NTX) and extended-release buprenorphine (XR-B) will participate in a randomized controlled trial throughout the state of Maryland, in which 240 incarcerated men and women will be randomly assigned within gender within jail to one of two arms: Arm 1. XR-B (n=120). XR-B in jail followed by 6 monthly injections post-release at a treatment program. Arm 2. XR-NTX (n=120). XR-NTX in jail, followed by 6 monthly injections post-release at a treatment program. In addition to the RCT the investigators will use a learning collaborative to examine the acceptability and feasibility of medications for opioid use disorder (MOUDs). Aim 1. To determine the effectiveness of XR-B compared to XR-NTX in terms of: Primary. (a) pharmacotherapy adherence (number of monthly injections received). Secondary. (b) illicit opioid urine test results; (c) self-reported illicit opioid use; (d) overdose events (non-fatal and fatal); (e) quality of life (i. physical health; ii. mental health); (f) HIV risk behaviors (i. sexual behavior; ii. needle use or sharing); and (g) criminal activity (i. crime days; ii. re-arrest; iii. re-incarceration). Aim 2. To use a learning collaborative involving all 7 RCT county jurisdictions as well as 3 additional counties that selected not to participate in the randomized trial to understand factors related to: (a) acceptability of providing long-acting agonists and antagonists in jail settings; and (b) feasibility of providing medication continuity of care from jail to community treatment providers. Aim 3. Calculate the cost to the correctional health system of implementing an XR-B or XR-NTX program, and determine the relative value of each strategy, including the costs associated with the subsequent interventions in the community, from a state-policymaker and societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female inmates at participating jails who are eligible for release within 120 days
* History of opioid use disorder (meeting DSM-5 criteria of moderate or severe opioid use disorder at the time of incarceration; individuals not meeting the opioid-disorder criterion will be eligible if they were treated in an opioid agonist treatment program during the year before incarceration)
* Suitability for XR-B and/or XR-NTX treatment as determined by medical evaluation
* Willingness to enroll in XR-B or XR-NTX treatment in jail
* Planning to live in one of the 7 participating counties and/or surrounding counties

Exclusion Criteria:

* Liver function test levels greater than 4 times normal;
* Active medical illness that may make participation hazardous (e.g., unstable diabetes, heart disease; moderate to severe renal impairment; adequately treated medical conditions are acceptable);
* Conditions or medications that may predispose to QTc prolongation (personal or family history of long QT syndrome, hypokalemia, medications that prolong QTc interval, e.g., macrolide antibiotics, azole antifungal compounds, anti-arrythmics, antipsychotics and antidepressant)
* Untreated psychiatric disorder that may make participation hazardous (e.g., untreated psychosis, bipolar disorder with mania; adequately treated psychiatric disorders and appropriate psychotropic medications will be allowed);
* History of allergic reaction to naltrexone and/or buprenorphine;
* Current chronic pain diagnosis for which opioids are prescribed;
* Pregnancy (for women);
* Breast-feeding (for women);
* Suicidal ideation (within the past 6 months);
* Body Mass Index (BMI) > 40;
* Inability to pass a study enrollment quiz;
* Currently enrolled in jail-based MOUD pharmacotherapy (methadone, buprenorphine, naltrexone)
* Enrolled in a methadone treatment program in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
pharmacotherapy adherence | 6-months post-release
  number of monthly injections received (0-6)

SECONDARY OUTCOMES:
illicit opioid urine screening test results | 1-7,12-months
  number of illicit opioid positive urine drug screen results
self-reported illicit opioid use | Baseline, 1-7,12-months
  self reported days of illicit opioid use
overdose events | Baseline, 1-7,12-months
  number of fatal and non-fatal overdoses
Patient-Reported Outcomes Measurement Information System | Baseline, 1-7,12-months
  physical, mental, and social health
  * scored 0: Death
  * scored < 1: A state worse than perfect health
Risk Assessment Battery (RAB) | Baseline, 1-7,12-months
  HIV risk behaviors; total score/40 (range=0-1)
Criminal activity | Baseline, 1-7,12-months
  number of days committed crime (20 crimes)
Re-arrest | 12-months
  time to rearrest (days to arrest)
Re-incarceration | 12-months
  time to re-incarceration (days to re-incarceration)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Gordon, DPA, Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086